CLINICAL TRIAL: NCT06408311
Title: A Safety and Tolerability Study of ENC=201-CED in Participants With Type 1 Diabetes Receiving Islet Infusion
Brief Title: Safety of ENC-201-CED ENCRT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Encellin (Industry)
Collaborators: resCON Research (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ENC201PD
Record Dates: First submitted 2024-05-02; First posted 2024-05-10 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism; Islet Infusion; Pancreas Transplant
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ENC-201-CED hPI (Experimental)
  Interventions: Combination Product: ENC-201-CED hPI

INTERVENTIONS:
Combination Product: ENC-201-CED hPI — macro-encapsulated human primary islets

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of ENC-201-CED in a subcutaneous space in patients with Type I diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Candidates must satisfy site's eligibility for standard of care islet infusion.

Exclusion Criteria:

* Candidates are excluded based on the site's criteria for standard of care islet infusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety | Day 1 through Day 134
  Rate of device-related Adverse Events (AE)

SECONDARY OUTCOMES:
Containment | post Day 120
  Assessment of number of islet equivalents (IEQ) in explants
Engraftment | post Day120
  Histopathology to examine degree of fibrosis (mm) from surface of CED.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Wei, PhD, Study Director — Encellin
Locations (2):
- Canada (2):
  - UHN, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No